CLINICAL TRIAL: NCT05609435
Title: Evaluating a Novel Follow-up Intervention to Improve the Delivery of Follow-up Care for Low-Risk Breast Cancer Survivors in Wisconsin
Brief Title: Intervention to Improve the Delivery of Follow-up Care for Low-Risk Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW22095; SMPH/SURGERY/SURG ONC (Other: UW Madison); Protocol Version 1/18/2024 (Other: UW Madison)
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: follow up care; low risk; health care delivery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a randomized, trial of REASSURE vs usual care within UW Health oncology clinics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REASSURE Follow Up care (Experimental)
  Interventions: Other: REASSURE
- Usual Follow Up Care (No Intervention)

INTERVENTIONS:
Other: REASSURE — REASSURE is comprised of three components that are intended to be integrated into survivorship care at each follow-up visit: 1) An online patient-reported outcome (PRO) assessment to comprehensively evaluate survivors' symptoms and concerns; 2) A tailored follow-up recommendation based on pre-established thresholds for reported symptoms and concerns. Survivors who report symptoms or concerns have a follow-up visit to discuss findings whereas survivors without symptoms or concerns will avoid a follow-up visit; and 3) Online survivorship messaging sent after the visit, which includes reassurance about the low recurrence risk, an overview of what to expect from follow-up, and steps survivors can take to reduce cancer risk.
  Arms: REASSURE Follow Up care

SUMMARY:
This study tests a novel intervention designed to optimize needed survivorship care for low-risk breast cancer survivors while reducing burdensome care with limited health benefits. This study examines whether the intervention, titled REASSURE, improves survivors' preparedness for survivorship. Up to 110 participants will be on study for up to 18 months.

DETAILED DESCRIPTION:
The investigators plan a single site prospective, randomized, trial that will compare the effect of REASSURE on survivor preparedness against usual care. Survivors will be identified from breast oncology clinics within UW Health.

REASSURE is comprised of three components: 1) the REASSURE PRO assessment, which assesses survivors' symptoms and/or concerns, 2) a recommendation for or against a follow-up visit based on survivors reported symptoms /concerns using pre-established thresholds, and 3) REASSURE survivorship messaging.

* Primary Objective

  * Compare survivors' preparedness for survivorship with REASSURE versus usual care.
* Secondary Objectives

  * Determine the acceptability of REASSURE for survivors living in rural and non-rural areas.
  * Assess changes in survivor reported symptoms and number of follow-up visits with REASSURE versus usual care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I, ER and/or PR positive, her2neu negative breast cancer within the last 6-24 monoths
* Willing to complete study procedures using email

Exclusion Criteria:

* Receipt of chemotherapy for the stage I ER and/or PR positive, her2neu negative breast cancer diagnosed within the last 6-24 months
* Participants will be excluded if they are unable to read and write in English or if, in the opinion of a treating clinician, have cognitive impairment that would prevent completion of study procedures
* Pregnancy, based on patient self-report. If a patient becomes pregnant during the study period, they will be removed from the study at that time.
* Diagnosis of a ER and PR negative, her2neu negative breast cancer or a her2neu positive breast cancer within the last 5 years

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Preparing for Life as a (New) Survivor (PLANS) Scale Score: Part 1 | up to 18 months
  Survivors' preparedness for survivorship will be assessed using Part 1 of the Preparing for Life as a (New) Survivor (PLANS) scale. This is an 11-item survey scored on a 4 point likert scale for a total possible range of score from 11 - 44 where higher scores indicate increased preparedness.
Preparing for Life as a (New) Survivor (PLANS) Scale Score: Part 2 | up to 18 months
  Survivors' confidence about follow-up will be assessed using Part 2 of the Preparing for Life as a (New) Survivor (PLANS) scale. This is a 5-item survey scored on a 10 point likert scale for a total possible range of score from 5 - 50 where higher scores indicate increased confidence.

SECONDARY OUTCOMES:
Number of Participants In Intervention Arm who would recommend this approach to follow-up to other survivors | up to 18 months
  REASSURE will be considered acceptable if ≥80% of survivors in the REASSURE arm respond "yes" to, "Would you recommend this approach to follow-up to other survivors?".
Number of Threshold-Level Symptoms Reported on the PRO Assessment | up to 18 months
  The number of threshold-level symptoms reported on the Patient Reported Outcome (PRO) assessment at each follow-up time point will be reported. This is based on the investigators' previously established thresholds of symptoms or concerns that warrant a visit. Some symptoms were "hard stops", meaning any reported symptom triggered a visit, other symptoms triggered a visit based on severity or level of interference.
Number of Threshold-Level Symptoms Survivors Perceive are Addressed on each visit | up to 18 months
Number of Follow Up Visits | up to 18 months
  The number of follow-up visits over the 18-month follow-up period will be counted. All follow-up visits that occur in medical oncology, radiation oncology, surgery, and survivorship clinics, including both physician and advanced practice provider visits will be counted.

OTHER OUTCOMES:
Number of Participants Who Received Recommended Cancer Care | up to 18 months
  Receipt of recommended cancer care over 18-months (chart review, yes/no)
Survivors' Experiences: Impact of Event Scale | up to 18 months
  Impact of Event Scale (measure of cancer-related anxiety) is a 15-item survey scored on a 5 point likert scale for a total possible range of scores from 15-75 where higher scores indicate higher anxiety.
Survivors' Experiences: Satisfaction with Information | up to 18 months
  Satisfaction with Information is measured using a 14-item survey scored on a 5 point likert scale for a total possible range of scores from 14-70 where higher scores indicate increased satisfaction with information.
Survivors' Experiences: Human Connection Scale Score | up to 18 months
  Human Connection Scale (measure of therapeutic alliance with providers) is a 10-item survey measured on a 5 point likert scale for a total possible range of scores from 10 to 50 where higher scores indicate higher connection with provider.
Survivors' Experiences: Quality of Follow Up Care | up to 18 months
  Quality of follow-up care using the question: "How would you rate the quality of follow-up care you received in the past 2 years?" This scored from 1 (poor) to 5 (excellent).
Healthcare Utilization: Number of Visits and Services Used | up to 18 months
  Healthcare utilization is measured via chart review, and includes use of ancillary services, visits with primary care, visits to urgent care/emergency room.
Healthcare Utilization: Number of MyChart Visits and Phone Calls | up to 18 months
  Healthcare utilization is measured via chart review, and includes number of my-chart visits and documented phone calls during 18 month study period.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Neuman, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Health Oncology Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No